CLINICAL TRIAL: NCT06940128
Title: Direct Ischemic Conditioning for Endovascular Recanalization for Anterior Large Vessel Occlusion (DICER-aLVO): a Prospective, Randomized, Open Label, Blinded-end Point, Phase 2, Multi-centre Study
Brief Title: Direct Ischemic Conditioning for Endovascular Recanalization for Anterior Large Vessel Occlusion (DICER-aLVO)
Acronym: DICER-aLVO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: General Hospital of Shenyang Military Region (Other)
Responsible Party: Principal Investigator, Hui-Sheng Chen, Director, General Hospital of Shenyang Military Region
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Y(2025)096
Record Dates: First submitted 2025-04-07; First posted 2025-04-23 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Ischemic Stroke
Keywords: Direct Ischemic Conditioning; stroke; Endovascular Recanalization
MeSH Terms: conditions — Ischemic Stroke; Stroke

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Direct Ischemic Conditioning Group A (Experimental): The protocol comprised 5 cycles of 30-s balloon inflations and 30-s deflations.
  Interventions: Procedure: Direct Ischemic Conditioning A
- Direct Ischemic Conditioning Group B (Experimental): The protocol comprised 4 cycles of 60-s balloon inflations and 60-s deflations.
  Interventions: Procedure: Direct Ischemic Conditioning B
- Direct Ischemic Conditioning Group C (Experimental): The protocol comprised 3 cycles of 120-s balloon inflations and 120-s deflations.
  Interventions: Procedure: Direct Ischemic Conditioning C
- Control group (No Intervention)

INTERVENTIONS:
Procedure: Direct Ischemic Conditioning A — Direct Ischemic Conditioning initiated within 5 minutes post-revascularization using either a balloon guiding catheter or a balloon catheter, positioned at the C1 segment of the ipsilateral internal carotid artery (ICA) to temporarily halt antegrade flow. The protocol comprised 5 cycles of 30-s balloon inflations and 30-s deflations.
  Arms: Direct Ischemic Conditioning Group A
Procedure: Direct Ischemic Conditioning B — Direct Ischemic Conditioning initiated within 5 minutes post-revascularization using either a balloon guiding catheter or a balloon catheter, positioned at the C1 segment of the ipsilateral internal carotid artery (ICA) to temporarily halt antegrade flow. The protocol comprised 4 cycles of 60-s balloon inflations and 60-s deflations.
  Arms: Direct Ischemic Conditioning Group B
Procedure: Direct Ischemic Conditioning C — Direct Ischemic Conditioning initiated within 5 minutes post-revascularization using either a balloon guiding catheter or a balloon catheter, positioned at the C1 segment of the ipsilateral internal carotid artery (ICA) to temporarily halt antegrade flow. The protocol comprised 3 cycles of 120-s balloon inflations and 120-s deflations.
  Arms: Direct Ischemic Conditioning Group C

SUMMARY:
Acute ischemic stroke (AIS) is the most common type of stroke, with high incidence rate and mortality. Endovascular therapy is currently the most effective treatment for AIS with large vessel occlusion, but only about 50% of patients achieve good outcome after endovascular therapy, while 50% of patients have poor prognosis, commonly referred to as ineffective perfusion. Therefore, how to improve ineffective perfusion is currently a hot topic.

Numerous studies have shown that Remote Ischemic Therapy (RIC) has a protective effect on ischemic stroke. Our recent RICAMIS study has demonstrated that RIC can significantly improve the functional prognosis of moderate acute ischemic stroke. Furthermore, direct ischemic conditioning has also showed neuroprotective effect. For example, in a rat model, within 2 minutes after reperfusion, using three cycles of 30 s reperfusion and 10 s occlusion for direct ischemic conditioning can effectively alleviate hyperperfusion and reduce cerebral infarction volume. Meanwhile, in previous clinical exploration studies, it was found that even induction by 5-minute ischemia and 5-minute reperfusion for up to 4 cycles is safe, feasible, and well tolerated for AIS patients receiving endovascular treatment. Immediate control of bilateral carotid artery blood flow after ischemia-reperfusion can significantly reduce cerebral infarction area and brain edema, and improve neurological function recovery in rats. Subsequent molecular mechanism studies have shown that direct ischemic conditioning can reduce the production of free radicals after cerebral ischemia-reperfusion, inhibit inflammatory reactions and cell apoptosis, downregulate the expression of signaling molecules mediating brain edema, promote Akt survival pathway, and improve the integrity of the blood-brain barrier, thereby exerting neuroprotective effects. Recent studies have also confirmed the safety and feasibility of direct ischemic conditioning for stroke patients achieving successful recanalization. More importantly, a recent cohort study has shown that direct ischemic conditioning can reduce infarct growth and brain edema after reperfusion in patients with AIS who have undergone thrombectomy for occlusion of large blood vessels in the anterior circulation, and improve prognosis after 90 days.

Based on the above discussion, this trial aims to evaluate the effectiveness and safety of direct ischemic conditioning for patients with AIS who have undergone thrombectomy for occlusion of large blood vessels in the anterior circulation.

ELIGIBILITY:
Inclusion Criteria:

-1. Over 18 years old; 2. The time from onset to randomization is less than 24 hours; 3. Patients with acute anterior artery occlusion and receiving successful recanalization (mTICI 2b-3) after endovascular treatment and with residual stenosis ≤ 50%; 4. Cerebral circulation time after successful recanalization: affected side ≤ healthy side; 5. PH2 hemorrhage was excluded by immediate postoperative CT examination; 6. Re-onset patients with first onset or past onset without sequelae such as limb paralysis should not affect the score of this NIHSS, and mRS Score of patients with past onset should be less than 2 points; 7. Signed informed consent by patient or their legally authorized representative.

Exclusion Criteria:

- 1. Spherical enlargement of the lesion site twice or more; 2. Proximal residual stenosis >50% for patients with tandem lesions; 3. Intracranial hemorrhagic diseases: cerebral hemorrhage, subarachnoid hemorrhage, etc.

4. Chronic liver disease, liver and kidney insufficiency, elevated ALT or AST (greater than 2 times the upper limit of normal), elevated serum creatinine (greater than 1.5 times the upper limit of normal) or dependent on kidney dialysis; 5. Women who are pregnant, have a pregnancy plan or are breastfeeding; 6. Combined with serious other diseases, life expectancy < 6 months; 7. Other conditions deemed inappropriate for participation in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-03-31 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with modified Rankin Score (mRS) 0 to 2 | at 90±7 days
  mRS ranges from 0-6, higher scores mean a worse outcome

SECONDARY OUTCOMES:
distribution of modified Rankin Score (mRS) | at 90±7 days
  mRS ranges from 0-6, higher scores mean a worse outcome
Proportion of patients with modified Rankin Score (mRS) 0 to 1 | at 90±7 days
  mRS ranges from 0-6, higher scores mean a worse outcome
Proportion of early neurological improvement | at 24 (-6/+24) hours
  early neurological improvement was defined as a 4 point or greater decrease in National Institute of Health stroke scale (NIHSS). NIHSS range from 0-42, higher scores mean a worse outcome
Change in National Institute of Health stroke scale (NIHSS) score | at 24 (-6/+24) hours
  NIHSS range from 0-42, higher scores mean a worse outcome
Change in National Institute of Health stroke scale (NIHSS) score | at 10±2 days
  NIHSS range from 0-42, higher scores mean a worse outcome
The amount of contrast exudation after treatment (CT assessment) | at 24 (-6/+24) hours
The amount of midline shift of the brain on neuroimaging after treatmet | at 24 (-6/+24) hours
Changes in brain circulation time after treatment (between healthy side and affected side, before and after treatment of affected side ischemia) | immediately after treatment
Recurrent stroke and new cardiovascular and cerebrovascular events | at 90±7 days
Proportion of balloon treatment-related complications (responsible vessel re-occlusion, vagal reflex, dissection, plaque shedding, and vasospasm during and after treatment) | immediately after treatment
Proportion of symptomatic intracranial hemorrhage | at 24 (-6/+24) hours
Proportion of occurrence of cerebral parenchymal hemorrhage types (PH1) and (PH2) | at 24 (-6/+24) hours
Proportion of serious adverse events | at 24 (-6/+24) hours
Proportion of all-cause deaths | at 10 days

OTHER OUTCOMES:
Changes in serum biomarkers | at 24 (-6/+24) hours
Changes in cerebral blood flow autoregulation ability | at 24 (-6/+24) hours

CONTACTS AND LOCATIONS:
Locations (1):
- General Hospital of Northern Theater Command, Shengyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: Undecided